CLINICAL TRIAL: NCT06998056
Title: A Phase 2, Open Label, 4-Week, Safety Study of Roflumilast Cream 0.05% Administered Once Daily in Infants Aged 3 Months to Less Than 2 Years With Atopic Dermatitis
Brief Title: Safety Study of Roflumilast Cream 0.05% in Infants Aged 3 Months to Less Than 2 Years With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-218
Record Dates: First submitted 2025-05-05; First posted 2025-05-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (Eczema)
Keywords: atopic dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Single arm open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 roflumilast cream 0.05% (open label) (Experimental): This single study arm is open label in which ARQ-151 cream 0.05% is applied daily for 4 weeks.
  Interventions: Drug: ARQ-151 cream 0.05%

INTERVENTIONS:
Drug: ARQ-151 cream 0.05% — ARQ-151 Cream 0.05% is applied once daily for 4 weeks in infants with atopic dermatitis (eczema).

SUMMARY:
This study will assess the safety and tolerability of ARQ-151 cream 0.05% applied once a day for 4 weeks in infants with atopic dermatitis (eczema).

DETAILED DESCRIPTION:
This study is an open label safety study in which ARQ-151 cream 0.05% is applied once a day for 4 weeks in infants with atopic dermatitis (eczema).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of a parent(s) or legal guardian(s), as required by local laws.
2. Males and females, ages 3 months to <2 years old at Day 1.
3. Diagnosed with mild to moderate Atopic Dermatitis (AD) for at least 1 month duration prior to or at the screening visit.
4. Has AD involvement of ≥3% BSA at Day1.
5. In good health as judged by the Investigator
6. Subjects and parent(s)/legal guardian(s) are considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects with any serious medical condition, clinically significant vital signs, or physical examination abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator.
2. Subjects who have unstable AD or any consistent requirement for high potency topical steroids to manage AD signs or symptoms.
3. Subjects previously treated with ARQ-151
4. Subjects currently undergoing allergy testing or food challenges, or plan to do so during the study.
5. Parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language. Subjects who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
6. Subjects who are family members of the clinical study staff or sponsor.

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events | 4 weeks
  Number of participants with adverse events during treatment will be assessed
Subject incidence of serious adverse events | 4 weeks
  Number of participants with serious adverse events during treatment will be assessed
Incidence of application site reactions | 4 weeks
  Number of subjects that experience an application site skin reaction by investigator assessment and application site reactions reported as adverse events will be assessed

CONTACTS AND LOCATIONS:
Locations (22):
- United States (17):
  - Arcutis Clinical Study Site 208, Birmingham, Alabama
  - Arcutis Clinical Study Site 221, Bryant, Arkansas
  - Arcutis Clinical Study Site 214, Fountain Valley, California
  - Arcutis Clinical Study Site 209, Rancho Santa Margarita, California
  - Arcutis Clinical Study Site 207, Coral Gables, Florida
  - Arcutis Clinical Study Site 217, Delray Beach, Florida
  - Arcutis Clinical Study Site 213, Jacksonville, Florida
  - Arcutis Clinical Study Site 223, Boise, Idaho
  - Arcutis Clinical Study Site 219, West Lafayette, Indiana
  - Arcutis Clinical Study Site 212, Minneapolis, Minnesota
  - Arcutis Clinical Study Site 211, Portsmouth, New Hampshire
  - Arcutis Clinical Study Site 220, Mason, Ohio
  - Arcutis Clinical Study Site 206, Portland, Oregon
  - Arcutis Clinical Study Site 222, Summerville, South Carolina
  - Arcutis Clinical Study Site 210, Bellaire, Texas
  - Arcutis Clinical Study Site 224, Fort Worth, Texas
  - Arcutis Clinical Study Site 202, San Antonio, Texas
- Canada (4):
  - Arcutis Clinical Study Site 203, Winnipeg, Manitoba
  - Arcutis Clinical Study Site 204, Halifax, Nova Scotia
  - Arcutis Clinical Study Site 216, Waterloo, Ontario
  - Arcutis Clinical Study Site 225, Saskatoon, Saskatchewan
- Arcutis Clinical Study Site 201, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Undecided